CLINICAL TRIAL: NCT01380548
Title: A Double-blind, Placebo Controlled Study to Assess Efficacy of 5-Aminolevulinic Acid in Subjects With Iron Deficiency Anemia
Brief Title: Effects of 5-Aminolevulinic Acid on Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: SBI ALApromo Co., Ltd., Japan (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: eki-396
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron; Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Iron alone (Placebo Comparator)
  Interventions: Dietary Supplement: Iron alone
- Low-dose 5-aminolevulinic acid (Experimental)
  Interventions: Dietary Supplement: Low-dose 5-aminolevulinic acid with iron
- Medium-dose 5-aminolevulinic acid (Experimental)
  Interventions: Dietary Supplement: Medium-dose 5-aminolevulinic acid with iron
- High-dose 5-aminolevulinic acid (Experimental)
  Interventions: Dietary Supplement: High-dose 5-aminolevulinic acid with iron

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo; once/day; for 12 weeks
  Arms: Placebo
Dietary Supplement: Iron alone — Iron (3 mg); once/day; for 12 weeks
  Arms: Iron alone
Dietary Supplement: Low-dose 5-aminolevulinic acid with iron — 5-Aminolevulinic acid (12.5 mg) and iron (3 mg); once/day; for 12 weeks
  Arms: Low-dose 5-aminolevulinic acid
Dietary Supplement: Medium-dose 5-aminolevulinic acid with iron — 5-Aminolevulinic acid (25 mg) and iron (3 mg); once/day; for 12 weeks
  Arms: Medium-dose 5-aminolevulinic acid
Dietary Supplement: High-dose 5-aminolevulinic acid with iron — 5-Aminolevulinic acid (50 mg) and iron (3 mg); once/day; for 12 weeks
  Arms: High-dose 5-aminolevulinic acid

SUMMARY:
This study is designed to evaluate efficacy and dose-dependency of 5-aminolevulinic acid in subjects with iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with hemoglobin ≥ 9.0 g/dl and ≤ 12.0 g/dl
* Willing not to donate blood during the study
* Informed consent signed

Exclusion Criteria:

* History of porphyria, hemochromatosis, or viral hepatitis
* Anemia other than iron deficiency
* BMI ≤ 18 kg/m2 or ≥ 30 kg/m2
* Pregnant or nursing a child
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease
* Subjects who are taking medicines or functional food that may affect hemoglobin level

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | Every 4 weeks (Overall 20 weeks)

SECONDARY OUTCOMES:
Serum ferritin level | Every 4 weeks (Overall 20 weeks)
Transferrin level | Every 4 weeks (Overall 20 weeks)
MCV level | Every 4 weeks (Overall 20 weeks)
TIBC level | Every 4 weeks (Overall 20 weeks)
Reticulocyte level | Every 4 weeks (Overall 20 weeks)
Red blood cell level | Every 4 weeks (Overall 20 weeks)
Hematocrit level | Every 4 weeks (Overall 20 weeks)
Serum iron level | Every 4 weeks (Overall 20 weeks)
Soluble transferrin receptor level | Week 0 (baseline) and Week 12
Hepcidin-25 level | Week 0 (baseline) and Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Japan